CLINICAL TRIAL: NCT02717572
Title: Reproducibility of 18F-FDG Uptake Measurements in Malignant Solid Tumors on PET/CT and PET/MR
Brief Title: 18F-FDG Uptake Measurements in Malignant Solid Tumors on PET/CT and PET/MR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201508093
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — Fluorodeoxyglucose F18; Positron-Emission Tomography; Tomography, X-Ray Computed; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- FDG-PET/CT and FDG-PET/MR (Experimental): * 10 mCI fludeoxyglucose IV bolus approximately 60 minutes before first PET/CT
  * Immediately following PET/CT scan, the participant will be moved to PET/MR scanner
  * The scans will take place at baseline and also one more time point between Day 1 and Day 7. There needs to be at least 24 hours between the baseline and repeat imaging
  Interventions: Radiation: Fludeoxyglucose F 18; Device: Positron Emission Tomography; Device: Computerized Tomography; Device: Magnetic Resonance Imaging

INTERVENTIONS:
Radiation: Fludeoxyglucose F 18
  Other Names: FDG; 18FDG
Device: Positron Emission Tomography
  Other Names: PET
Device: Computerized Tomography
  Other Names: CT; CAT
Device: Magnetic Resonance Imaging
  Other Names: MRI

SUMMARY:
In the current study, the investigators plan to expand the knowledge of Positron Emission Tomography/Magnetic Resonance (PET/MR) reliability by assessing the repeatability of fludeoxyglucose (FDG) standardized uptake values (SUV) measurements, as well as apparent diffusion coefficients (ADC) measurements, in a broad population of patients with malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed malignant solid tumors (local or metastatic, newly diagnosed or recurrent disease).
* Patient must have at least one lesion measuring ≥ 2.0 cm.
* 18 years of age or older.
* Ability to provide informed consent.

Exclusion Criteria:

* Cancer therapy within 30 days of baseline imaging.
* Uncontrolled intercurrent illness including, but not limited to active infections.
* Patients with insulin-dependent diabetes.
* Patients with metal devices in the body including, but not limited to metallic joint prostheses, artificial heart valves, pacemakers, and cochlear implants.
* Patients who are pregnant or nursing.
* Inability to tolerate 60 minutes of PET imaging.
* Inability to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-06-05 (Actual)

PRIMARY OUTCOMES:
Variability of repeated quantitative measures of FDG uptake as measured by SUVmax | Completion of study (up to Day 7)
  -SUVmax is the maximum standardized uptake value (SUV) of the area of showing metabolic activity and this is used to show response
Variability of repeated quantitative measures of FDG uptake as measured by SUVpeak | Completion of study (up to Day 7)
  -SUVpeak, which is defined as the average SUV within a 1 cubic cm volume within the region of the tumor with the highest metabolic activity
Repeatability of diffusion-weighted imaging on PET/MR as measured by difference in mean ADC | Completion of study (up to Day 7)
  * DW MRI is a method of mapping the diffusion process of water within and between tissues
  * Water diffusion is described quantitatively by apparent diffusion coefficients (ADC)
Repeatability of diffusion-weighted imaging on PET/MR as measured by differences in minimum ADC | Completion of study (up to Day 7)
  * DW MRI is a method of mapping the diffusion process of water within and between tissues
  * Water diffusion is described quantitatively by apparent diffusion coefficients (ADC)

SECONDARY OUTCOMES:
Evaluation of the ratio of SUVmax and ADCmin | Completion of study (up to Day 7)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Wahl, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu